CLINICAL TRIAL: NCT06656182
Title: Effect of SNAGs and Scapular Mobilizations in Patients With Scapulocostal Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/MS-PT/01941 Rabia Asif
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Scapulocostal Syndrome
Keywords: non specific neck pain; SNAGs; Scapular mobilizations; NDI

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical and Thoracic SNAGs (Experimental): Cervical and Thoracic SNAGs with 6 reps and 1 set along with cervical and shoulder muscle stretching and scapular mobilizations
  Interventions: Other: Cervical and Thoracic SNAGs
- traditional physical therapy and scapular mobilizations (Active Comparator): cervical and shoulder muscle stretching and scapular mobilizations
  Interventions: Other: traditional physical therapy and scapular mobilizations

INTERVENTIONS:
Other: Cervical and Thoracic SNAGs — cervical SNAGs (C3-C7) and thoracic SNAGs (T1-T12) with 6 repetitions of 1 set three times per week for 4 weeks along with scapular mobilizations of 10 repetitions of 1 set and stretching of trapezius (upper, middle and lower fibers), levator scapulae and rhomboids (major and minor)
  Arms: Cervical and Thoracic SNAGs
Other: traditional physical therapy and scapular mobilizations — scapular mobilizations of 10 repetitions of 1 set and stretching of trapezius (upper, middle and lower fibers), levator scapulae and rhomboids (major and minor)
  Arms: traditional physical therapy and scapular mobilizations

SUMMARY:
To determine the impact of SNAGs and Scapular mobilizations on pain, cervical and shoulder Range of motion and functional outcomes in individuals with Scapulocostal Syndrome.

DETAILED DESCRIPTION:
The rationale for employing SNAGS (Sustained Natural Apophyseal Glides) in treating scapulocostal syndrome is multifaceted. By targeting specific joint surfaces and soft tissue structures, SNAGS aim to address joint dysfunction, alleviate pain, and improve mobility in the scapulothoracic region. These sustained gliding movements not only modulate pain signals but also promote relaxation and reduce muscle tension, thereby enhancing the effectiveness of therapeutic exercises aimed at strengthening the surrounding musculature. Additionally, SNAGS facilitate proper muscle activation patterns, optimizing muscle function and coordination. Their adaptability allows for a patient-centered approach, ensuring tailored treatment that considers individual symptoms, mobility deficits, and treatment goals, ultimately promoting better functional outcomes in individuals with scapulocostal syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age- 18 to 40 years.

  * Male and female both
  * Nonspecific neck pain with a duration of greater than 3 months
  * No pain reproduction on isometric muscle testing in shoulder.
  * Patients who could not achieve 60 degrees of upward rotation when elevating the arms above the head i.e. presence of scapular dyskinesia
  * pain with a referral pattern while receiving manual pressure of at least 3 points on the medial scapular muscles (levator scapulae, rhomboid major, rhomboid minor, and serratus posterior superior) evaluated through Travels and Simon criteria.
  * Discomfort, pain, or limitations in neck extension, neck rotation bilaterally, shoulder forward flexion, shoulder abduction attributed to SCS.
  * Willing to provide informed consent to participate in the study.

Exclusion Criteria:

* Musculoskeletal pathologies affecting the cervical spine or lower extremities (e.g., herniated disc, cervical radiculopathy, cervical stenosis, shoulder labral tear).

  * history of degenerative shoulder joint disease
  * rotator cuff dysfunction
  * Thoracic outlet syndrome
  * Brachial neuralgia
  * shoulder impingement syndrome
  * adhesive capsulitis
  * Pregnant individuals due to potential discomfort.
  * Open wounds, infections, or skin conditions at pain site.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Neck disability index | 4th week
  changes from baseline The Neck Disability Index (NDI) serves as a valuable tool for evaluating neck pain issues, drawing on the framework of the Oswestry index for back pain and the Pain Disability Index. Its effectiveness lies in its focus on the impact of neck pain on daily activities, reflecting the specific concerns and experiences of individual patients.
  Comprising 10 sections, each containing 5 questions related to affected activities, the index allows patients to select the response that best represents their situation, with scores ranging from 0 to 5.

SECONDARY OUTCOMES:
NPRS | every week
  changes from baseline Pain through NPRS at the end of every week for 4 weeks
Cervical and Shoulder ROM | every week
  changes from baseline at the end of every week till last week

CONTACTS AND LOCATIONS:
Overall Officials: Asmar Fatima, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- DSK physio and Rehab Center, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No